CLINICAL TRIAL: NCT05870644
Title: Acute Effects of Exercise at Different Temperatures on Nasal Blood Flow and Symptoms in Patient With Allergic Rhinitis.
Brief Title: Acute Effects of Exercise at Different Temperatures in Allergic Rhinitis Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Wannaporn Tongtako, Ph.D., Principal investigator, Chulalongkorn University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EX PHYSIO SPSC 6
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Allergic Rhinitis
Keywords: aerobic exercise; allergic rhinitis; nasal blood flow; peak nasal inspiratory flow; acute exercise
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: Fifteen patients with allergic rhinitis aged between 18 and 35 years who had a positive skin prick test to house dust mite (D. pteronyssinus). The experiment was a crossover design in which each participant was given aerobic exercise by ergometer in two difference temperatures room : 25 degree celsius and 34 degree celsius. Rhinitis symptoms, nasal blood flow, heart rate, and oxygen saturation were measured before, during exercise at 15, 30, and 45 minutes, and after exercise at 0, 15 and 30 minutes in each temperature. Moreover, blood pressure, peak nasal inspiratory flow, pulmonary functions, respiratory muscle strength, and fractional exhaled nitric oxide were measured before and after exercise at 0, 15 and 30 minutes in each temperature.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise in room temperature at 25 degree Celsius. (Experimental): The participants received a moderate exercise program of cycling at moderate intensity (50-60% HRR) for 60 minutes in room temperature at 25 degree Celsius.
  Interventions: Other: Cycling exercise in room temperature at 25 degree Celsius.
- Exercise in room temperature at 34 degree Celsius. (Experimental): The participants received a moderate exercise program of cycling at moderate intensity (50-60% HRR) for 60 minutes in room temperature at 34 degree Celsius.
  Interventions: Other: Cycling exercise in room temperature at 34 degree Celsius.

INTERVENTIONS:
Other: Cycling exercise in room temperature at 25 degree Celsius. — The participants received a aerobic exercise of cycling for 60 minutes in room temperature at 25 degree Celsius.
  Arms: Exercise in room temperature at 25 degree Celsius.
Other: Cycling exercise in room temperature at 34 degree Celsius. — The participants received a aerobic exercise of cycling for 60 minutes in room temperature at 34 degree Celsius.
  Arms: Exercise in room temperature at 34 degree Celsius.

SUMMARY:
The purpose of this study was to determine the effects of exercise at different temperatures on nasal blood flow and symptoms in allergic rhinitis patients.

DETAILED DESCRIPTION:
Fifteen patients with allergic rhinitis aged between 18 and 35 years who had a positive skin prick test to house dust mite (D. pteronyssinus). The experiment was a crossover design in which each participant was given aerobic exercise by ergometer in two difference temperatures room : 25 degree celsius and 34 degree celsius. Rhinitis symptoms, nasal blood flow, heart rate, and oxygen saturation were measured before, during exercise at 15, 30, and 45 minutes, and after exercise at 0, 15 and 30 minutes in each temperature. Moreover, blood pressure, peak nasal inspiratory flow, pulmonary functions, respiratory muscle strength, and fractional exhaled nitric oxide were measured before and after exercise at 0, 15 and 30 minutes in each temperature.

ELIGIBILITY:
Inclusion Criteria:

* Subjects had a clinical history of persistent rhinitis, and had positive skin prick test to house dust mite (D. pteronyssinus)
* Persistent allergic rhinitis
* Subjects with known asthma, chronic rhinosinusitis, Lung cancer and Emphysema diseases were excluded.
* BMI 18.5 - 24.9 kg/m2
* Subjects will ask to abstain from taking antihistamine for at least 5 days, leukotriene receptor antagonist for at least 1 week, and nasal steroids for at least 2 weeks prior to the start of the experiment.
* Subjects will ask to abstain from taking any form of dietary supplement during the experiment.
* Subjects had no exercise training program (not exercise regularly or not exercise for 30 minutes or more at least 3 times per week during the past 6 months)

Exclusion Criteria:

* Accident that are unable to continue the research, such as accidental injury or illness, etc.
* Participants did not voluntarily participate.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
Rhinitis symptom scores change | Change among before, during exercise at 15, 30, and 45 minutes, and after exercise at 0, 15 and 30 minutes in each temperature.
  Nasal symptoms were assessed using Total Nasal Symptom Score (TNSS) questionnaire. The subjects were asked to score symptoms of persistent allergic rhinitis before, during exercise at 15, 30, and 45 minutes, and after exercise at 0, 15 and 30 minutes in each temperature. The total nasal symptom scores were computed as the sum of four individual nasal symptom scores; nasal congestion, itching, sneezing, and rhinorrhea. The scores ranged from 0 to 3 scale (0=none, 1=mild, 2=moderate, 3= severe)
Nasal blood flow change | Change among before, during exercise at 15, 30, and 45 minutes, and after exercise at 0, 15 and 30 minutes in each temperature.
  Laser Doppler flowmetry (DRT4 moor instrument, UK.) was used to measure of the nasal blood flow (NBF). A lateral endoscopic probe with a flexible nylon sheath 1.34-mm-diameter flexible nylon sheath was placed to the front of the nose. Nasal blood flow measurements were performed before, during exercise at 15, 30, and 45 minutes, and after exercise at 0, 15 and 30 minutes in each temperature.
Peak nasal inspiratory flow change | Change before and after exercise at 0, 15 and 30 minutes in each temperature.
  he subjects placed a mask, which is turned onto a plastic cylinder through which the air passes during inspiration, over the nose and mouth and inspired forcefully through the nose, with lips tightly closed. Inside the cylinder, there is a diaphragm that moves to the airflow, and the maximum peak flow is registered in a scale range from 30-370 L/min. During the procedure, the subjects placed a mask over the nose and mouth and inspired forcefully through the nose, with lips tightly closed.

SECONDARY OUTCOMES:
Fractional exhaled nitric oxide | Change before and after exercise at 0, 15 and 30 minutes in each temperature.
  Participants inhaled deeply for two to three seconds before exhaling slowly. Normally, it took 10 seconds to exhale.
Pulmonary functions change | Change before and after exercise at 0, 15 and 30 minutes in each temperature.
  The participants were asked to wear a nose clip while sitting on a chair, and the researcher gave the participants the step-by-step protocol to prevent an incorrect maneuver. For the FVC maneuver, three cycles of slow normal breathing were performed before demonstrating forced inspiration and expiration.
Respiratory muscle strength change | Change before and after exercise at 0, 15 and 30 minutes in each temperature.
  Respiratory muscle strength was assessed by measuring Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP) in cmH2O. The participants were in a sitting position using a portable handheld mouth pressure meter (i.e., MicroRPM) with a nose clip. For the MIP measurement, the participants were asked to exhale until they felt no air remaining in their lungs (starting with the functional residual capacity [FRC] point), then held the device on their mouth and inhaled forcefully for 1-2 seconds. For the MEP measurement, the participants were asked to inhale until their lungs were completely filled with air (starting with the total lung capacity [TLC] point), then they kept the device on their mouth and exhaled forcefully for 1-2 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sports Science, Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brozek JL, Bousquet J, Agache I, Agarwal A, Bachert C, Bosnic-Anticevich S, Brignardello-Petersen R, Canonica GW, Casale T, Chavannes NH, Correia de Sousa J, Cruz AA, Cuello-Garcia CA, Demoly P, Dykewicz M, Etxeandia-Ikobaltzeta I, Florez ID, Fokkens W, Fonseca J, Hellings PW, Klimek L, Kowalski S, Kuna P, Laisaar KT, Larenas-Linnemann DE, Lodrup Carlsen KC, Manning PJ, Meltzer E, Mullol J, Muraro A, O'Hehir R, Ohta K, Panzner P, Papadopoulos N, Park HS, Passalacqua G, Pawankar R, Price D, Riva JJ, Roldan Y, Ryan D, Sadeghirad B, Samolinski B, Schmid-Grendelmeier P, Sheikh A, Togias A, Valero A, Valiulis A, Valovirta E, Ventresca M, Wallace D, Waserman S, Wickman M, Wiercioch W, Yepes-Nunez JJ, Zhang L, Zhang Y, Zidarn M, Zuberbier T, Schunemann HJ. Allergic Rhinitis and its Impact on Asthma (ARIA) guidelines-2016 revision. J Allergy Clin Immunol. 2017 Oct;140(4):950-958. doi: 10.1016/j.jaci.2017.03.050. Epub 2017 Jun 8. PMID 28602936
- [Background] Min YG. The pathophysiology, diagnosis and treatment of allergic rhinitis. Allergy Asthma Immunol Res. 2010 Apr;2(2):65-76. doi: 10.4168/aair.2010.2.2.65. Epub 2010 Mar 24. PMID 20358020
- [Background] Katel P, Pinkaew B, Talek K, Tantilipikorn P. Pattern of Aeroallergen Sensitization and Quality of Life in Adult Thai Patients With Allergic Rhinitis. Front Allergy. 2021 Nov 15;2:695055. doi: 10.3389/falgy.2021.695055. eCollection 2021. PMID 35387043
- [Background] Olsson P, Bende M. Influence of environmental temperature on human nasal mucosa. Ann Otol Rhinol Laryngol. 1985 Mar-Apr;94(2 Pt 1):153-5. doi: 10.1177/000348948509400211. PMID 3994233
- [Background] Bailey RS, Casey KP, Pawar SS, Garcia GJ. Correlation of Nasal Mucosal Temperature With Subjective Nasal Patency in Healthy Individuals. JAMA Facial Plast Surg. 2017 Jan 1;19(1):46-52. doi: 10.1001/jamafacial.2016.1445. PMID 27918749